CLINICAL TRIAL: NCT04775576
Title: Comparison of Conventional Fluid Management Protocol With Targeted Pleth Variability Index (PVI) Monitoring Protocol During Total Abdominal Hysterectomy and Bilateral Salpingooferectomy Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ummahan Dalkilinc Hokenek, Anesthesiology and Reanimation Specialist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020/514/172/4
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Intraoperative Hypotension; Intraoperative Complications; Hypervolemia; Acute Renal Failure; Perioperative/Postoperative Complications; Volume Overload
MeSH Terms: conditions — Intraoperative Complications; Edema; Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): This group will have fluid theraphy due to conventional methods. The participants in this group will have 8-10 ml/kg/hour cristalloid infusion. If the mean arterial pressure (MAP) is <65 mmHg or the decrease in MAP is more than 20%, 250 ml iv colloid will be applied. If the decrease in MAP continues despite the colloid bolus or if the MAP is below 65 mmHg, noradrenaline infusion will be started.
  Interventions: Other: Conventional fluid theraphy; Other: Anesthesia method
- Group 2 (Active Comparator): Patients in the PVI group will be started on maintenance fluid therapy at 2-3 ml / kg / hour. In addition to standard monitoring, if PVI is <13% and OAB≥65mmHg in measurements made with PVI, current fluid therapy will continue. If PVI is <13% and MAP <65 mmHg, noradrenaline infusion will be started. If PVI is> 13% and OAB≥65 mmHg, 250 ml iv colloid bolus will be administered, and iv colloid bolus will be continued until the PVI is <13% in the 5-minute follow-ups. If PVI> 13% and MAP <65 mmHg, patients should receive 250 ml i.v. colloid infusion will be given, if MAP <65mmHg continues in 5 minutes follow-up, 250 ml i.v. Colloid and noradrenaline infusion will be started and repeated until the OAB≥65 mmHg and PVI <13%.
  Interventions: Other: Pleth Variability Index; Other: Anesthesia method

INTERVENTIONS:
Other: Pleth Variability Index — Conventional fluid management is widely used in clinical practice. In this method, the fluid need of the patient is decided according to pulse, arterial blood pressure, central venous pressure, urine output and clinical condition. In the targeted fluid therapy method, besides static parameters such as pulse, arterial blood pressure, central venous pressure; Dynamic parameters such as Stroke volume variability (SVV), pulse pressure variability (PPV), pleth variability index (PVI), continuous hemoglobin (SpHb) are also used noninvasively.
  Arms: Group 2
Other: Conventional fluid theraphy — 8-10 ml / kg / hour iv fluid maintenance will be started for the control group. If the mean arterial pressure (MAP) is <65 mmHg or the decrease in MAP is more than 20%, 250 ml iv colloid will be applied. If the decrease in MAP continues despite the colloid bolus or if the MAP is below 65 mmHg, noradrenaline infusion will be started.
  Arms: Group 1
Other: Anesthesia method — All patients included in the study will be premedicated with 1mg of midazolam after monitoring with pulse, non-invasive blood pressure, oxygen saturation. Then, invasive arterial cannulation will be applied and continuous blood pressure monitoring will be done. In the PVI group, non-invasive PVI and SpHb monitoring will also be performed from the other upper extremity without arterial cannulation. After two minutes of preoxygenation, anesthesia induction will be started. Anesthesia induction doses used routinely in our clinic include iv 2 mg / kg propofol, 0.6 mg / kg rocuronium and 2 μg / kg fentanyl. Sevoflurane will be administered by inhalation during anesthesia maintenance after tracheal intubation.

SUMMARY:
This study aims to compare the volume management methods performed by using conventional method and PVI monitoring in intraoperative fluid treatment during bilateral salpingo-oophorectomy and total hysterectomy operation.

DETAILED DESCRIPTION:
Intraoperative fluid management is very important in terms of postoperative organ perfusion and complications. While various complications such as acute renal failure, hypotension, arrhythmia, anastomotic leakage can be seen due to intraoperative hypovolemia; Hypervolemia can cause pulmonary edema, postoperative pneumonia, prolonged mechanical ventilation need, delayed wound healing, gastrointestinal system (GIS) edema and decreased intestinal motility.

Increasing the quality of intraoperative fluid therapy is a situation that may affect the morbidity and mortality of patients due to all these reasons.

Conventional fluid management is widely used in clinical practice. In this method, the fluid need of the patient is decided according to pulse, arterial blood pressure, central venous pressure, urine output and clinical condition. In the targeted fluid therapy method, besides static parameters such as pulse, arterial blood pressure, central venous pressure; Dynamic parameters such as Stroke volume variability (SVV), pulse pressure variability (PPV), pleth variability index (PVI), continuous hemoglobin (SpHb) are also used noninvasively. Studies related to SpHb, which provides noninvasive continuous hemoglobin monitoring in accordance with pulse oximetry, show that there is a decrease in blood product transfusion compared to cases managed with conventional laboratory follow-up.

Our primary goal is to compare the control group (conventional fluid management) with the PVI group (Pleth Variability Index and SpHb guided targeted fluid management) protocol.

For this purpose, we aim to compare the amount of crystalloids and blood products, blood lactate, serum creatinine and electrolyte levels applied in the intraoperative period as a result of both protocols. Our secondary aim will be to compare the length of stay in the hospital.

The study is planned as a single center, prospective, randomized controlled clinical study. It was aimed to evaluate fluid therapy during elective total abdominal hysterectomy and bilateral salpingooferectomy operation. Before the operation, patients will be divided into 2 groups randomly. For randomization, the automatic system on the randomization.com website will be used. All patients included in the study will be premedicated with 1mg of midazolam after monitoring with pulse, non-invasive blood pressure, oxygen saturation. Then, invasive arterial cannulation will be applied and continuous blood pressure monitoring will be done. In the PVI group, non-invasive PVI and SpHb monitoring will also be performed from the other upper extremity without arterial cannulation. After two minutes of preoxygenation, anesthesia induction will be started. Anesthesia induction doses used routinely in our clinic include iv 2 mg / kg propofol, 0.6 mg / kg rocuronium and 2 μg / kg fentanyl. Sevoflurane will be administered by inhalation during anesthesia maintenance after tracheal intubation. Initially, all patients will be given 250 ml intravenous crystalloid. Then 8-10 ml / kg / hour iv fluid maintenance will be started for the control group. If the mean arterial pressure (MAP) is <65 mmHg or the decrease in MAP is more than 20%, 250 ml iv colloid will be applied. If the decrease in MAP continues despite the colloid bolus or if the MAP is below 65 mmHg, noradrenaline infusion will be started. Patients in the PVI group will be started on maintenance fluid therapy at 2-3 ml / kg / hour. In addition to standard monitoring, if PVI is <13% and OAB≥65mmHg in measurements made with PVI, current fluid therapy will continue. If PVI is <13% and MAP <65 mmHg, noradrenaline infusion will be started. If PVI is> 13% and OAB≥65 mmHg, 250 ml iv colloid bolus will be administered, and iv colloid bolus will be continued until the PVI is <13% in the 5-minute follow-ups. If PVI> 13% and MAP <65 mmHg, patients should receive 250 ml i.v. colloid infusion will be given, if MAP <65mmHg continues in 5 minutes follow-up, 250 ml i.v. Colloid and noradrenaline infusion will be started and repeated until the OAB≥65 mmHg and PVI <13%. The decision to transfuse in both groups will be taken under the guidance of the European Society of Anesthesia (ESA) perioperative bleeding management guidelines. In the control group, hemorrhage will be monitored with laboratory Hb values, while SpHb and laboratory Hb values will be evaluated together in the PVI group.

Patients in the ASA1-2-3 risk group who will undergo elective total abdominal hysterectomy and bilateral salpingo-oophorectomy under general anesthesia, between the ages of 18-65, will be included in this study. The study will be conducted with 80 people.

In both groups, continuous arterial blood pressure, heart rate, oxygen saturation and arterial blood gas, lactate concentration at hourly intervals, hemoglobin, hematocrit, serum urea, creatinine, sodium, potassium, chlorine values, hospital stay, hourly intervals, intraoperative hourly and postoperatively 24 hours later, The amount of crystalloids and blood products used intraoperatively, postoperative volume dependent complications and their frequency will be evaluated.

The study will be conducted by anesthesiologists in the operating rooms located in the central campus of our hospital.

ELIGIBILITY:
Inclusion Criteria:

Total abdominal hysterectomy and bilateral salpingooferectomy operation is planned Patients in the ASA 1-2-3 group

Exclusion Criteria:

Under 18 years old Severe cardiac arrhythmia Ejection fraction ≤ 30% Acute and / or chronic renal failure Patients who need more than 8ml / kg tidal volume due to advanced stage COPD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — total abdominal hysterectomy and bilateral salpingooferectomy operation
Enrollment: 78 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
compare the control group (conventional fluid management) with the PVI group (Pleth Variability Index and SpHb guided targeted fluid management) protocol. | 0-180 minute
  compare the amount of crystalloids,colloids and blood products, blood lactate, serum creatinine and electrolyte levels applied in the intraoperative period as a result of both protocols.

SECONDARY OUTCOMES:
Postoperative length of stay in hospital | 24 hours
  Evaluation of postoperative hospital stay in both groups
Postoperative kidney injury | 24 hours
  Present of postoperative kidney injury/failure
Postoperative Lung complications | 24 hours
  Present of hypervolemia related lung edema

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lutfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Holte K, Sharrock NE, Kehlet H. Pathophysiology and clinical implications of perioperative fluid excess. Br J Anaesth. 2002 Oct;89(4):622-32. doi: 10.1093/bja/aef220. No abstract available. PMID 12393365
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Background] Raikhel M. Accuracy of noninvasive and invasive point-of-care total blood hemoglobin measurement in an outpatient setting. Postgrad Med. 2012 Jul;124(4):250-5. doi: 10.3810/pgm.2012.07.2584. PMID 22913913
- [Background] Miller RD, Ward TA, Shiboski SC, Cohen NH. A comparison of three methods of hemoglobin monitoring in patients undergoing spine surgery. Anesth Analg. 2011 Apr;112(4):858-63. doi: 10.1213/ANE.0b013e31820eecd1. Epub 2011 Mar 8. PMID 21385985
- [Result] Doherty M, Buggy DJ. Intraoperative fluids: how much is too much? Br J Anaesth. 2012 Jul;109(1):69-79. doi: 10.1093/bja/aes171. Epub 2012 Jun 1. PMID 22661747
- [Result] Arieff AI. Fatal postoperative pulmonary edema: pathogenesis and literature review. Chest. 1999 May;115(5):1371-7. doi: 10.1378/chest.115.5.1371. PMID 10334155